CLINICAL TRIAL: NCT03839368
Title: Stability of Angle Fracture Fixation With (K) Shaped Titanium Miniplates Versus Two Conventional Miniplates: Randomized Clinical Trial
Brief Title: Stability of Angle Fracture Fixation With (K) Shaped Titanium Miniplates Versus Two Miniplates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Mahmoud Ahmed Mohamed, Resident of Oral and Maxillofacial Surgery - Nasser Institute Hospital for research & treatment / Master Candidate of Oral & Maxillofacial surgery, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-02-03
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-04

CONDITIONS: Mandible Fracture
Keywords: angle fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant
Masking Description: Cards will have sequential numbers one number for each card then these cards will be placed within opaque sealed envelopes. Then these envelops will be placed in a container (box), each participant will grasp one envelope the day of procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K plate (Experimental): fixation of angle fracture using K plate versus two miniplates
  Interventions: Procedure: fixation of angle fracture
- Conventional two miniplates (Active Comparator): fixation of angle fracture using K plate versus two miniplates
  Interventions: Procedure: fixation of angle fracture

INTERVENTIONS:
Procedure: fixation of angle fracture — open reduction and internal fixation of angle fracture

SUMMARY:
In patients with angle fracture , will the (K) shaped titanium miniplates provide more stable fixation than two conventional miniplates? Many studies have been conducted to compare between different techniques of fixation used in angle fracture fixation. The driving force behind this study was to design a new plate that would overcome the disadvantages of the other plating techniques but has the advantages & simplicity of the Champy technique (simple intraoral approach and few major complications). This new miniplate gives more biomechanical stability than the conventional Champy plate. More over the placement of a 3D miniplate or two separate miniplates for fixing angle fractures is more difficult and mostly will require a transbuccal approach , with increased surgical trauma, longer operation time unlike the new plate that could provide the clinician with a simple and reliable solution.

DETAILED DESCRIPTION:
In the past two decades, rigid internal fixation with miniplate has become the standard treatment modality in the management of mandibular fracture.

The optimal management of mandibular angle fractures remains controversial, thus continuous experimental & clinical studies are being conducted to determine the best miniplate design which will provide the best postoperative stability & resistance to mechanical function.

Since Michelet et al.& Champy et al. recommended the use of a single (4-6 holes) monocortical plate , it become an acceptable method for angle fractures fixation.

Several surgeons have documented low complication rates with (Champy technique).But, according to the most recent experimental & clinical studies, the stability provided by the miniplate fixation has become a point of debate among surgeons.Many researchers have argued that internal fixation with a passive miniplate along the external oblique line, following Champy's ideal osteosynthesis line principle, produces a tension effect that may yield a failure of osteosynthesis & gap at inferior border of the mandible.And that pushed researches to conduct more studies to evaluate many plate & screw systems and even suggest new designs for better stable postoperative results.

In 2014, B.T.Suer et al, designed a new noncompression 3D miniplates , basically it has one straight section and two lateral extensions. The straight section of this new design, which has four holes, was adapted to the superior border of the external oblique ridge & provides similar advantages to the Champy technique (an intraoral approach, a single miniplate, & the use of monocortical screws) .And the two lateral extensions, with one hole each, were then bent over to adapt to the buccal cortex of the ascending ramus along the external oblique ridge to resist lateral & torsional forces.

Fresh, frozen cadavers of 15 healthy sheep were obtained for this study, sheep were used in this study owing to the similarities in size & thickness to the human mandible. All of the mandibles were stripped of their soft tissues & sectioned through the midline, between the central incisors. 30 hemimandibles were randomly divided into two groups , these groups were then fixed with two different plating techniques (the new design & one conventional miniplates). And they were all examined for stability and resistance to mechanical forces (vertical, lateral, or tensile).

The driving force behind this study was to design a new plate that would overcome the disadvantages of the other plating techniques but has the advantages & simplicity of the Champy technique (simple intraoral approach and few major complications). This new miniplate gives more biomechanical stability than the conventional Champy plate. These findings are correlated to those of in vitro biomechanical study done by Alkan et al. that showed that Champy technique has less favourable biomechanical behaviour than biplanar fixation and 3D strut plate. In addition the new plate provide greater stability when subjected to lateral displacing forces.

More over the placement of a 3D miniplate or two separate miniplates for fixing angle fractures is more difficult and mostly will require a transbuccal approach , with increased surgical trauma, longer operation time unlike the new plate that could provide the clinician with a simple and reliable solution.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral angle fracture.
2. Patients free from any systemic disease & bone metabolism diseases.
3. No sex predilection
4. Age range ( 15-70)

Exclusion Criteria:

1. Comminuted fragmented & infected angle fractures.
2. Bilateral angle fracture.
3. Systemic diseases.
4. bone metabolism diseases

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-04-11 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Stability of angle fracture fixation | 3 months
  Inter-ramus distance (fixed position at the lingual), inter-mental distance will be obtained from the immediate postoperative facial bone CT & after 3 months. Comparison between the 2 records will be done to assess the stability of fixation technique.
  Bone density will be measured by Hounsfield unit at fracture site immediate postoperative & after 3 months using F.B.CT.

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Mohamed, BDS, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suer BT, Kocyigit ID, Kaman S, Tuz HH, Tekin U, Atil F. Biomechanical evaluation of a new design titanium miniplate for the treatment of mandibular angle fractures. Int J Oral Maxillofac Surg. 2014 Jul;43(7):841-5. doi: 10.1016/j.ijom.2014.01.011. Epub 2014 Feb 24. PMID 24582290
- [Derived] El-Sherif HM, Ali S, Talaat M, Mubarak F. Stability and Clinical Outcomes of Angle Fracture Fixation Using Sagittal Split Plate (SSOP) Versus Two Miniplates: Randomized Clinical Trial. J Maxillofac Oral Surg. 2024 Feb;23(1):107-113. doi: 10.1007/s12663-022-01817-z. Epub 2022 Nov 16. PMID 38312972